CLINICAL TRIAL: NCT04193917
Title: Confounding Factors in Ocular Surface Microbiome Research
Acronym: CoFa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S63155
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-07

CONDITIONS: Ocular Surface Microbiome
Keywords: Ocular surface microbiome; Temporal stability; Confounding factors

STUDY DESIGN:
Intervention Model Description: A conjunctival swab will be taken from healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- conjunctival swab (Other): A conjunctival swab of both eyes will be taken
  Interventions: Diagnostic Test: Conjunctival swab

INTERVENTIONS:
Diagnostic Test: Conjunctival swab — A conjunctival swab of both eyes will be taken at the same time together with an extensive questionnaire.

SUMMARY:
To elucidate confounding factors in ocular surface microbiome research and to confirm the presence of a core ocular surface microbiome and its temporal stability.

DETAILED DESCRIPTION:
The investigator will take a conjunctival sample of both eyes of a group of volunteers together with an extensive questionnaire. Furthermore, 50 volunteers will be sampled repeatedly during one year or two years.

ELIGIBILITY:
Inclusion Criteria:

* The subject is fluent in written and verbal Dutch
* The subject is capable of giving informed consent

Exclusion Criteria:

* Use of glaucoma drops
* Use of antibiotic drops < 1 month before sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2019-11-24 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Richness and evenness of distribution of the microbial flora measured as operational taxonomic units on a single moment | 20 minutes for samples and filling the questionnaires
  A conjunctival swab and extensive questionnaire will be taken to search for a core ocular surface microbiome and confounding factors
Change in richness and evenness of distribution of the microbial flora, measured as operational taxonomic units, over time | 20 minutes for the first sample and questionnaire, 5 minutes for all other visits
  A conjunctival swab will be taken on different points in time to investigate the temporal stability of the conjunctival microbial flora

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Delbeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Department of Ophthalmology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided